CLINICAL TRIAL: NCT04282109
Title: Phase II Multicenter Randomized Trial to Assess the Efficacy and Safety of First Line Nivolumab in Combination With Paclitaxel in Subjects With R/M HNSCC Unable for Cisplatin-based Chemotherapy (NIVOTAX)
Brief Title: Study to Assess the Efficacy and Safety of Nivolumab in Combination With Paclitaxel in Subjects With Head and Neck Cancer Unable for Cisplatin-based Chemotherapy (NIVOTAX)
Acronym: NIVOTAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Collaborators: Bristol-Myers Squibb (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2019-01/CA209-7HE; 2019-002922-60 (EudraCT Number)
Record Dates: First submitted 2020-02-12; First posted 2020-02-24 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; Squamous cell carcinoma; Nivolumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Nivolumab; Paclitaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): NIVOTAX (nivolumab + paclitaxel, follow by maintenance with nivolumab)
  Interventions: Drug: Nivolumab + Paclitaxel
- Arm 2 (Active Comparator): ERBITAX (cetuximab + paclitaxel, follow by maintenance with cetuximab)
  Interventions: Drug: Cetuximab + Paclitaxel

INTERVENTIONS:
Drug: Nivolumab + Paclitaxel — Combination treatment: Nivolumab 240 mg will be administered via IV infusion every 2 weeks. Paclitaxel 80mg/m2 will be administered via IV infusion weekly. After 12 weeks from the start of the combined treatment paclitaxel will be stopped.
  Maintenance treatment with nivolumab 480 mg every 4 weeks will start two weeks after the last administration of nivolumab 240 mg. Once nivolumab is administered at 480 mg, paclitaxel can no longer be administered.
  Nivolumab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
  Arms: Arm 1
Drug: Cetuximab + Paclitaxel — Combination treatment: Cetuximab 250 mg/m2 (first dose of 400 mg/m2) administered via IV infusion weekly plus weekly paclitaxel (80 mg/m2) administered via IV infusion.
  After 12 weeks from the start of the combined treatment paclitaxel will be stopped and weekly cetuximab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
  Arms: Arm 2

SUMMARY:
Chemotherapy for recurrent or metastatic head and neck squamous cell carcinoma is palliative and usually platinum based, and the patients often present with poor physical condition. Consequently, many of them are not able to withstand a platinum-based chemotherapy. The addition of taxanes to the armamentarium of drugs improve the outcome in this group of patients. An alternative and better tolerated regimen for these patients is paclitaxel in combination with cetuximab, included the in guidelines of the Spanish Society of Medical Oncology.

Recently, new treatments such as immune-checkpoint inhibitors have shown promising activity and good tolerability in patients with recurrent or metastatic head and neck squamous cell carcinoma and has been included in the recently published guidelines from the Society for Immunotherapy of Cancer. Nivolumab (anti-PD1) has been approved for patients progressing on or after platinum-based therapy, as it clearly impacts on overall survival.

This randomized phase II study will evaluate the efficacy of nivolumab plus paclitaxel for first-line treatment of recurrent or metastatic HNSCC in the platinum ineligible and platinum refractory settings. Control arm will be paclitaxel in combination with cetuximab, treatment included in the guidelines of the Spanish Society of Medical Oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care.
2. Histologically confirmed HNSCC (oral cavity, oropharynx, hypopharynx, larynx) not amenable to therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
3. Patients not previously treated for recurrent/metastatic disease.
4. Radiographically measurable disease as defined by RECIST version 1.1. Previously irradiated lesions can only be considered as measurable disease if disease progression according to RECIST version 1.1.
5. Patients unable for cisplatin-based chemotherapy, defined "unable" by:

   1. Karnofsky 70% or
   2. Karnofsky 80-100% and amenable to chemotherapy, but:

   i. Impaired renal function, creatinine clearance >30 mL/min and <80 mL/min GFR could be assessed by direct measurement (EDTA or creatinine clearance) if available or by calculation from serum or plasma creatinine (see annex 5), or

   ii. grade ≥2 hearing loss, according to the NCI CTCAE v 5.0, or

   iii. Class III heart failure according to the New York Heart Association (annex 9), or

   iv. History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds or

   v. Prior dose of cisplatin ≥225 mg/m² for locally advanced disease (a patient who received prior RT + 3 cycles of cisplatin 100 mg/m2 or 3 cycles induction TPF (with cisplatin ≥75/m2) for locally advanced primary HN cancer can be included), or

   vi. Disease progression or relapse during or within 6 months of receiving platinum-based therapy administered as neoadjuvant, adjuvant therapy or as concomitant chemotherapy with radiotherapy and have received at least 200 mg/m2 of cisplatin.
6. Male or female patients aged ≥18 years. Patients aged ≥70 years old can only be included with a G8 (Geriatric 8) health status screening score ≥ 14.
7. Clinical laboratory values as specified below within 28 days before the first dose of study drug:

   1. Total bilirubin must be ≤2 × the upper limit of normal (ULN).
   2. Magnesium ≥ lower limit of normal.
   3. Calcium ≥ lower limit of normal.
   4. ALT and AST must be ≤3 × ULN unless liver metastases are present, in which case they must be ≤5x ULN.
   5. Hemoglobin must be ≥9 g/dL, absolute neutrophil count (ANC) must be ≥1.500/µL, WBC must be ≥2.000/µL and platelet count must be ≥100.000/µL.
8. Subjects who have received radiation as primary therapy are eligible if radiation therapy treatment was completed > 4 weeks prior to inclusion.
9. Documentation of PD-L1 status by IHC performed by the central lab at randomization. A pre-treatment tumor tissue sample should be sent. A newly obtained biopsy (within 6 months prior to start of study treatment) is preferred but an archival sample is acceptable, if several tumor samples are available, testing should be performed on the most recently obtained tumor sample.
10. Documentation of HPV p16 status (OPC) is required for HNSCC tumor of the oropharynx. For subjects with oropharyngeal cancer, sites are defined in annex 8. HPV status of tumor tissue has to be locally determined at screening by any of the following methods: p16 IHC, in situ hybridization, or polymerase chain reaction based assay. If HPV status by p16 IHC is positive result confirmation by PCR is mandatory.

Exclusion Criteria:

1. Male or female patients aged <18 years. Patients aged ≥ 70 years old should not be included with a G8 (Geriatric 8) health status screening score < 14.
2. Karnofsky <70%.
3. Patients that meets more than one of the following criteria:

   1. Karnofsky 70%,
   2. Impaired renal function, creatinine clearance >30 mL/min and <80 mL/min GFR could be assessed by direct measurement (EDTA or creatinine clearance) if available or by calculation from serum or plasma creatinine (see annex 5),
   3. Class III heart failure according to the New York Heart Association (annex 9).
4. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy except for alopecia, vitiligo, hear loss and the laboratory values defined in the inclusion criteria.
5. Histologically confirmed recurrent or metastatic squamous cell carcinoma of unknown primary, of the nasopharynx or non-squamous histologies (eg, mucosal melanoma).
6. Active brain metastases or leptomeningeal metastases.
7. Carcinomatous meningitis.
8. Active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or unexpected conditions of recurrence in the absence of an external trigger are allowed to be included.
9. Diagnosis of immunodeficiency or any condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of treatment.
10. History of pneumonitis requiring treatment with steroids; history of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest CT scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
11. Patients with a history of interstitial lung disease cannot be included if they have symptomatic ILD (Grade 3-4) and/or poor lung function.
12. Prior therapy with experimental antitumor vaccines; any T-cell co-stimulation agents or inhibitors of checkpoint pathways, such as anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody; or other agents specifically targeting T cells are prohibited.
13. Any serious medical or psychiatric illness, including drug or alcohol abuse, that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
14. Life-threatening illness unrelated to cancer.
15. Female patients who are lactating and breast-feeding or a positive serum pregnancy test during the screening period.
16. Systemic anticancer treatment or radiotherapy less than 4 weeks or 5 half-lives, whichever is longer, before the first dose of study treatment or not recovered from acute toxic effects from prior chemotherapy and radiotherapy.
17. Prior treatment with investigational agents ≤21 days (≤4 weeks for monoclonal antibodies with evidence of PD) or ≤5 their half-lives (whichever is shorter) before the first dose of study treatment. A minimum of 10 days should elapse from prior therapy to initiating protocol therapy.
18. Major surgery within 14 days before the first dose of study drug and not recovered fully from any complications from surgery.
19. Systemic infection requiring IV antibiotic therapy or other serious infection within 14 days before the first dose of study drug.
20. Known human immunodeficiency virus (HIV) positive (testing not required), or known acquired immunodeficiency syndrome (AIDS).
21. Patients with positive test for hepatitis B virus or hepatitis C virus indicating presence of virus, eg, Hepatitis B surface antigen (HBsAg) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).
22. Active secondary malignancy that requires treatment. Patients with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required during the study period
23. Any clinically significant co-morbidities, such as uncontrolled pulmonary disease, known impaired cardiac function or clinically significant cardiac disease, active central nervous system disease, active infection, or any other condition that could compromise the patient's participation in the study.
24. Patients with history of hypersensitivity reactions to study drugs (nivolumab, cetuximab or paclitaxel) or any of their excipients.
25. Symptomatic peripheral neuropathy of Grade ≥ 2 based on the CTCAE v5.0
26. Pulmonary embolism, deep vein thrombosis, or other significant thromboembolic event ≤ 8 weeks prior to starting the study treatment.
27. History of severe skin disorder that in the opinion of the investigator may interfere with study conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Mesia, MD, Principal Investigator — Hospital Universitari Germans Trias i Pujol de Badalona; Lara Iglesias, MD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (21):
- Spain (21):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Donostia- Donostia Unibertsitate Ospitalea, San Sebastián, San Sebastían
  - Centro Oncoloxico de Galicia, A Coruña
  - Hospital Universitari Germans Trias i Pujol de Badalona, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Institut Català D´Oncologia- Hospital Duran i Reynals, Barcelona
  - Hospital Universitari de Girona Dr. Josep, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico la Fe, Valencia
  - Hospital Clínico Universitario Lozano, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: NIVOTAX (nivolumab + paclitaxel, follow by maintenance with nivolumab)
  Nivolumab + Paclitaxel: Combination treatment: Nivolumab 240 mg will be administered via IV infusion every 2 weeks. Paclitaxel 80mg/m2 will be administered via IV infusion weekly. After 12 weeks from the start of the combined treatment paclitaxel will be stopped.
  Maintenance treatment with nivolumab 480 mg every 4 weeks will start two weeks after the last administration of nivolumab 240 mg. Once nivolumab is administered at 480 mg, paclitaxel can no longer be administered.
  Nivolumab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
- Arm 2: ERBITAX (cetuximab + paclitaxel, follow by maintenance with cetuximab)
  Cetuximab + Paclitaxel: Combination treatment: Cetuximab 250 mg/m2 (first dose of 400 mg/m2) administered via IV infusion weekly plus weekly paclitaxel (80 mg/m2) administered via IV infusion.
  After 12 weeks from the start of the combined treatment paclitaxel will be stopped and weekly cetuximab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 93 | 48
Completed | 93 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: NIVOTAX (nivolumab + paclitaxel, follow by maintenance with nivolumab).
  Nivolumab + Paclitaxel: Combination treatment: Nivolumab 240 mg will be administered via IV infusion every 2 weeks. Paclitaxel 80mg/m2 will be administered via IV infusion weekly. After 12 weeks from the start of the combined treatment paclitaxel will be stopped.
  Maintenance treatment with nivolumab 480 mg every 4 weeks will start two weeks after the last administration of nivolumab 240 mg. Once nivolumab is administered at 480 mg, paclitaxel can no longer be administered.
  Nivolumab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
- Arm 2: ERBITAX (cetuximab + paclitaxel, follow by maintenance with cetuximab).
  Cetuximab + Paclitaxel: Combination treatment: Cetuximab 250 mg/m2 (first dose of 400 mg/m2) administered via IV infusion weekly plus weekly paclitaxel (80 mg/m2) administered via IV infusion.
  After 12 weeks from the start of the combined treatment paclitaxel will be stopped and weekly cetuximab will be continued alone until disease progression, unacceptable toxicity or withdrawal of consent up to a maximum of 24 months.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 93 | 48 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 27 | 69
  >=65 years | 51 | 21 | 72
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66.8 [59 to 75] | 64 [57 to 70.5] | 65.9 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 73 | 36 | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 93 | 47 | 140
  Arab | 0 | 1 | 1
Smoking habits: Has the patient ever smoked? [Count of Participants; unit: Participants]
  Yes | 75 | 11 | 86
  No | 18 | 37 | 55
Metastatic disease at diagnosis [Count of Participants; unit: Participants]
  Yes | 8 | 3 | 11
  No | 85 | 45 | 130
Karnofsky performance status [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment.
  70%= Care for self. Unable to carry on normal activity or to do active work 80%= Normal activity with effort 90%=Able to carry on normal activities. Minor signs or symptoms of disease 100%= Normal, no complaints
  Participants
    70% | 36 | 16 | 52
    80-100% | 57 | 32 | 89
PD-L1 CPS [Count of Participants; unit: Participants] — PD-L1 positive = ≥ 1 CPS A positive CPS for PD-L1 determination means that the test result indicates detectable PD-L1 expression on tumour cells and/or immune cells within the tumour microenvironment. A higher CPS is usually associated with a higher likelihood of response to immunotherapy.
  PD-L1 negative = <1 CPS
  A negative PD-L1 result based on the CPS (Combined Positive Score) means there is little to no expression of PD-L1 in the tumor sample, which may limit the effectiveness or eligibility for certain immunotherapy treatments, depending on the cancer type and clinical guidelines.
  Participants
    <1 | 20 | 11 | 31
    ≥1 | 73 | 37 | 110
Type of disease [Count of Participants; unit: Participants]
  Loco-regional disease | 40 | 27 | 67
  Loco-regional disease + M1 | 26 | 12 | 38
  Metastatic disease | 27 | 9 | 36
Unable platinum [Count of Participants; unit: Participants]
  Platinum-refractory | 25 | 13 | 38
  Cumulative cisplatin dose ≥ 225 mg/m² | 15 | 8 | 23
  Platinum sensitive but unable | 53 | 27 | 80
Smoking habits: Does the patient currently smoke? [Count of Participants; unit: Participants]
  Yes | 21 | 9 | 30
  No | 72 | 39 | 111
Alcohol consumption [Count of Participants; unit: Participants]
  No | 31 | 20 | 51
  Current | 14 | 12 | 26
  Former | 41 | 15 | 56
  Unknown | 7 | 1 | 8
Primary tumor location [Count of Participants; unit: Participants]
  Oral cavity | 32 | 18 | 50
  Oropharynx | 33 | 14 | 47
  Larynx | 17 | 5 | 22
  Hypopharynx | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Two Years Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death. For subjects without documentation of death, OS will be censored on the last date the subject was known to be alive.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 24.7 [15.9 to 33.5] | 13.4 [3.6 to 23.2]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of first documented disease progression, as assessed by the investigator using RECIST 1.1 criteria, or death due to any cause, whichever occurs first.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
months | 5.6 [3.5 to 7.6] | 5.3 [2.7 to 7.9]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the number of subjects with a best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized subjects for each treatment group.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 37.6 [27.8 to 47.5] | 37.5 [23.8 to 51.2]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) is defined as the number of subjects with a best overall response (BOR) of a complete response (CR), partial response (PR) or stable disease (SD) divided by the number of randomized subjects for each treatment group.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 74.2 [65.3 to 83.1] | 79.2 [67.7 to 90.7]

5. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) is defined as the time between the date of first confirmed response to the date of the first documented tumor progression (per RECIST 1.1), or death due to any cause, whichever occurs first.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 35 | 18
month | 9 [7.6 to 10.5] | 7.6 [4.9 to 10.4]

6. Secondary Outcome: 6-months Progression-free Survival Rate
Description: Probability of progression at 6 months.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 47.5 [37.3 to 57.7] | 50.0 [35.9 to 64.1]

7. Secondary Outcome: Overall Survival in Patients ≥ 70 Years.
Description: OS is defined as the time between the date of randomization and the date of death.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 37 | 13
months | 13.03 [3.9 to 22.2] | 14.54 [7.99 to 21.01]

8. Secondary Outcome: Progression Free Survival in Patients ≥ 70 Years.
Description: as for outcome 2
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 37 | 13
month | 6.48 [2.22 to 10.73] | 9.97 [3.59 to 16.34]

9. Secondary Outcome: Overall Response Rate in Patients ≥ 70 Years.
Description: as for outcome 3
Time Frame: Up to 2 years
Population: Patients ≥ 70 years.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 37 | 13
percentage of participants | 40.5 | 53.8

10. Secondary Outcome: Overall Survival Based on PDL1 Expression (CPS).
Description: OS is defined as the time between the date of randomization and the date of death.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1 - CPS <1: NIVOTAX - CPS <1
- Arm 1 - CPS >=1: NIVOTAX - CPS >=1
- Arm 2 - CPS <1: ERBITAX - CPS <1
- Arm 2 - CPS >=1: ERBITAX - CPS >=1
Arm/Group | Arm 1 - CPS <1 | Arm 1 - CPS >=1 | Arm 2 - CPS <1 | Arm 2 - CPS >=1
Number analyzed (Participants) | 20 | 73 | 11 | 37
months | 11.94 [8.55 to 15.33] | 12.24 [8.90 to 15.57] | 14.54 [7.51 to 21.57] | 11.18 [8.99 to 13.38]

11. Secondary Outcome: Progression Free Survival Based on PDL1 Expression (CPS).
Description: as for outcome 2
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 - CPS <1 | Arm 1 - CPS >=1 | Arm 2 - CPS <1 | Arm 2 - CPS >=1
Number analyzed (Participants) | 20 | 73 | 11 | 37
months | 7.6 [0.55 to 14.65] | 5.56 [4.16 to 6.95] | 8.72 [2.65 to 14.79] | 5.33 [2.94 to 7.71]

12. Secondary Outcome: Overall Response Rate Based on PDL1 Expression (CPS).
Description: as for outcome 3
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - CPS <1 | Arm 1 - CPS >=1 | Arm 2 - CPS <1 | Arm 2 - CPS >=1
Number analyzed (Participants) | 20 | 73 | 11 | 37
percentage of participants | 45.0 | 35.6 | 27.3 | 40.5

13. Secondary Outcome: Overall Survival Based on Cisplatin Ineligibility.
Description: OS is defined as the time between the date of randomization and the date of death.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1 - Group 1: NIVOTAX - Group 1
  Platinum resistant population:
  - Patients who have experienced disease progression or relapse during or within 6 months of receiving platinum-based therapy administered as neoadjuvant, adjuvant therapy or as concomitant chemotherapy with radiotherapy and have received at least 200 mg/m2 of cisplatin.
- Arm 1 - Group 2: NIVOTAX - Group 2
  Platinum sensitive but unable for cisplatin based therapy according to one of these criteria:
  1. Karnofsky grade 70% or
  2. Impaired renal function, creatinine clearance >30 mL/min and <80 mL/min GFR could be assessed by direct measurement (EDTA or creatinine clearance) if available or by calculation from serum or plasma creatinine, or
  3. Class III heart failure according to the New York Heart Association, or
  4. Grade ≥2 hearing loss, according to the NCI CTCAE v 5.0, or
  5. History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds.
- Arm 1 - Group 3: NIVOTAX - Group 3
  Platinum sensitive but prior dose of cisplatin ≥225 mg/m² for locally advanced disease (one third of the patients - 47 patients) (a patient who received prior RT + 3 cycles of cisplatin 100 mg/m2 or 3 cycles induction TPF (with cisplatin ≥75/m2) for locally advanced primary HN cancer). The interval from the last cycle of cisplatin and the start of first line treatment for R/M disease is >6 months.
- Arm 2 - Group 1: ERBITAX - Group 1
  Platinum resistant population:
  - Patients who have experienced disease progression or relapse during or within 6 months of receiving platinum-based therapy administered as neoadjuvant, adjuvant therapy or as concomitant chemotherapy with radiotherapy and have received at least 200 mg/m2 of cisplatin.
- Arm 2 - Group 2: ERBITAX - Group 2
  Platinum sensitive but unable for cisplatin based therapy according to one of these criteria:
  1. Karnofsky grade 70% or
  2. Impaired renal function, creatinine clearance >30 mL/min and <80 mL/min GFR could be assessed by direct measurement (EDTA or creatinine clearance) if available or by calculation from serum or plasma creatinine, or
  3. Class III heart failure according to the New York Heart Association, or
  4. Grade ≥2 hearing loss, according to the NCI CTCAE v 5.0, or
  5. History of allergic reactions to cisplatin, carboplatin, or other platinum-containing compounds.
- Arm 2 - Group 3: ERBITAX - Group 3
  Platinum sensitive but prior dose of cisplatin ≥225 mg/m² for locally advanced disease (one third of the patients - 47 patients) (a patient who received prior RT + 3 cycles of cisplatin 100 mg/m2 or 3 cycles induction TPF (with cisplatin ≥75/m2) for locally advanced primary HN cancer). The interval from the last cycle of cisplatin and the start of first line treatment for R/M disease is >6 months.
Arm/Group | Arm 1 - Group 1 | Arm 1 - Group 2 | Arm 1 - Group 3 | Arm 2 - Group 1 | Arm 2 - Group 2 | Arm 2 - Group 3
Number analyzed (Participants) | 25 | 53 | 15 | 13 | 27 | 8
months | 8.95 [2.08 to 15.82] | 14.14 [11.39 to 16.90] | 10.49 [6.55 to 14.44] | 7.5 [4.83 to 10.16] | 14.54 [8.85 to 20.23] | 12.14 [7.7 to 16.61]

14. Secondary Outcome: Progression Free Survival Based on Cisplatin Ineligibility.
Description: as for outcome 2
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 - Group 1 | Arm 1 - Group 2 | Arm 1 - Group 3 | Arm 2 - Group 1 | Arm 2 - Group 2 | Arm 2 - Group 3
Number analyzed (Participants) | 25 | 53 | 15 | 13 | 27 | 8
months | 4.84 [0.11 to 9.56] | 5.56 [3.02 to 8.1] | 10.23 [6.63 to 16.83] | 2.53 [1.78 to 3.24] | 7.53 [6.64 to 8.43] | 8.26 [6.8 to 9.71]

15. Secondary Outcome: Overall Response Rate Based on Cisplatin Ineligibility.
Description: as for outcome 3
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - Group 1 | Arm 1 - Group 2 | Arm 1 - Group 3 | Arm 2 - Group 1 | Arm 2 - Group 2 | Arm 2 - Group 3
Number analyzed (Participants) | 25 | 53 | 15 | 13 | 27 | 8
percentage of participants | 32.0 | 39.6 | 40.0 | 15.4 | 51.9 | 25.0

16. Secondary Outcome: Overall Survival Based on Karnofsky.
Description: OS is defined as the time between the date of randomization and the date of death.
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm 1 - Karnofsky-PS 70%: NIVOTAX - Karnofsky-PS 70%
- Arm 1 - Karnofsky-PS 80-100%: NIVOTAX - Karnofsky-PS 80-100%
- Arm 2 - Karnofsky-PS 70%: ERBITAX - Karnofsky-PS 70%
- Arm 2 - Karnofsky-PS 80-100%: ERBITAX - Karnofsky-PS 80-100%
Arm/Group | Arm 1 - Karnofsky-PS 70% | Arm 1 - Karnofsky-PS 80-100% | Arm 2 - Karnofsky-PS 70% | Arm 2 - Karnofsky-PS 80-100%
Number analyzed (Participants) | 35 | 57 | 16 | 32
months | 13.03 [10.04 to 16.01] | 11.32 [6.45 to 16.19] | 11.18 [6.48 to 15.89] | 12.14 [10.68 to 13.59]

17. Secondary Outcome: Progression Free Survival Based on Karnofsky.
Description: as for outcome 2
Time Frame: Up to 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 - Karnofsky-PS 70% | Arm 1 - Karnofsky-PS 80-100% | Arm 2 - Karnofsky-PS 70% | Arm 2 - Karnofsky-PS 80-100%
Number analyzed (Participants) | 35 | 57 | 16 | 32
months | 6.48 [3.39 to 9.56] | 5.56 [4.2 to 6.92] | 4.84 [3.80 to 5.87] | 7.07 [3.38 to 10.76]

18. Secondary Outcome: Overall Response Rate Based on Karnofsky.
Description: as for outcome 3
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - Karnofsky-PS 70% | Arm 1 - Karnofsky-PS 80-100% | Arm 2 - Karnofsky-PS 70% | Arm 2 - Karnofsky-PS 80-100%
Number analyzed (Participants) | 36 | 57 | 16 | 32
percentage of participants | 41.6 | 35.1 | 43.7 | 34.4

19. Secondary Outcome: Percentage of Patients With AEs
Description: Percentage of patients with AEs in relation with total number of treated patients
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 100 | 100

20. Secondary Outcome: Percentage of Patients With Grade 3 and Grade 4 AEs
Description: Percentage of patients with Grade 3 and Grade 4 AEs in relation with total number of treated patients
Time Frame: 2 years
Population: Patients with at least one adverse event G≥3 during study
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 72.0 | 68.8

21. Secondary Outcome: Percentage of Patients With SAEs
Description: Percentage of patients with SAEs in relation with total number of treated patients
Time Frame: Up to 45 months
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 93 | 48
percentage of participants | 57.0 | 54.2

22. Secondary Outcome: Percentage of Patients Who Discontinued Due to AEs
Description: Percentage of patients who discontinued due to AEs in relation with total number of treated patients
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Groups:
- Arm 1 - Combination Phase: NIVOTAX - Combination phase
- Arm 1 - Monotherapy Phase: NIVOTAX - Monotherapy phase
- Arm 2 - Combination Phase: ERBITAX - Combination phase
- Arm 2 - Monotherapy Phase: ERBITAX - Monotherapy phase
Arm/Group | Arm 1 - Combination Phase | Arm 1 - Monotherapy Phase | Arm 2 - Combination Phase | Arm 2 - Monotherapy Phase
Number analyzed (Participants) | 93 | 59 | 48 | 33
percentage of participants | 14.0 | 10.2 | 10.4 | 6.1

ADVERSE EVENTS:
Time Frame: Up to 45 months
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 79/93 | 43/48
Serious Adverse Events (participants affected / at risk) | 53/93 | 26/48
Other Adverse Events (participants affected / at risk) | 93/93 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=93) | Arm 2 (N=48)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Gastrostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Product dispensing error (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 7 (8) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Submaxillary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1)
Hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (9) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6)
Sepsis (Infections and infestations) | 3 (3) | 1 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stoma site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=93) | Arm 2 (N=48)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 1 (2)
Hypertension (Vascular disorders) | 5 (7) | 1 (1)
Asthenia (General disorders) | 57 (166) | 29 (61)
Crepitations (General disorders) | 0 (0) | 4 (5)
Fatigue (General disorders) | 11 (22) | 3 (7)
Mucosal inflammation (General disorders) | 15 (32) | 16 (42)
Oedema peripheral (General disorders) | 5 (6) | 3 (4)
Pain (General disorders) | 9 (10) | 4 (8)
Pyrexia (General disorders) | 15 (22) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7) | 0 (0)
Amylase increased (Investigations) | 5 (10) | 1 (1)
Lipase increased (Investigations) | 6 (15) | 2 (3)
Neutrophil count decreased (Investigations) | 4 (9) | 4 (6)
Dizziness (Nervous system disorders) | 6 (8) | 4 (4)
Headache (Nervous system disorders) | 8 (10) | 2 (4)
Neuropathy peripheral (Nervous system disorders) | 10 (14) | 7 (15)
Neurotoxicity (Nervous system disorders) | 22 (38) | 10 (16)
Paraesthesia (Nervous system disorders) | 6 (8) | 5 (5)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 41 (86) | 19 (47)
Neutropenia (Blood and lymphatic system disorders) | 17 (37) | 11 (18)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (5)
Cheilitis (Gastrointestinal disorders) | 2 (3) | 4 (7)
Constipation (Gastrointestinal disorders) | 23 (29) | 14 (16)
Diarrhoea (Gastrointestinal disorders) | 26 (40) | 14 (24)
Dry mouth (Gastrointestinal disorders) | 5 (7) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 16 (19) | 8 (8)
Nausea (Gastrointestinal disorders) | 13 (15) | 6 (6)
Odynophagia (Gastrointestinal disorders) | 9 (11) | 5 (7)
Vomiting (Gastrointestinal disorders) | 9 (11) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (36) | 6 (8)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (9)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (18) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 10 (13) | 25 (58)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (9)
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (14)
Hypothyroidism (Endocrine disorders) | 13 (17) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (20) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 11 (13) | 3 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 6 (7)
COVID-19 (Infections and infestations) | 3 (3) | 3 (3)
Oral candidiasis (Infections and infestations) | 5 (7) | 2 (2)
Paronychia (Infections and infestations) | 1 (1) | 5 (8)
Pneumonia (Infections and infestations) | 5 (6) | 0 (0)
Respiratory tract infection (Infections and infestations) | 16 (24) | 7 (11)
Urinary tract infection (Infections and infestations) | 9 (9) | 4 (6)
Decreased appetite (Metabolism and nutrition disorders) | 17 (35) | 14 (17)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8) | 15 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT04282109/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT04282109/SAP_001.pdf